CLINICAL TRIAL: NCT03702062
Title: Dynamic Prediction of Heart Failure Using Real-time Functional Status and Electronic Health Record Data in the Ambulatory Setting
Brief Title: Dynamic Heart Failure Prediction With Real-time Functional Status Data in the Ambulatory Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HF1
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Arm (Experimental): Participants will be asked to measure self-assessed 6 minute walk test via the smart phone application twice a week for 2 months after discharge from a heart failure hospitalization, and weekly thereafter for 6 months.
  Interventions: Diagnostic Test: 6 Minute Walk Test Smart phone Application

INTERVENTIONS:
Diagnostic Test: 6 Minute Walk Test Smart phone Application — The intervention requests participants to user the smart phone application at prescribed frequencies during the follow-up period.

SUMMARY:
Heart failure is the number one cause of hospital readmission in those over 65 years of age and the current standard-of-care of weight self-monitoring is inadequate to predict exacerbation. This project aims to improve the monitoring of heart failure disease progression through the use of real-time, up-to-date data obtained both from a smart phone-based tool and from the electronic health record. The goal is to develop a low-risk, clinically validated method to estimate dynamic heart failure risk to enable the provision of earlier, more effective outpatient interventions that decrease hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for decompensated heart failure
* Age >=18 years
* Owns a smart phone
* Willing to measure self assess 6 minute walk test weekly

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-21 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization | 12 months
  hospital inpatient admission or emergency room visit

SECONDARY OUTCOMES:
Heart failure mortality | 12 months
  Death from heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Tison, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided